CLINICAL TRIAL: NCT03092427
Title: Evaluation of the Effectiveness of a Probiotic Treatment on Clinical Activity, Relapse Rates and Modification of the Intestinal Microbiota in Patients With Juvenile Idiopathic Arthritis (JIA)
Brief Title: Probiotic Treatment in Juvenile Idiopathic Arthritis (JIA)
Acronym: PERMAJI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P150934
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic VSL#3 (Experimental)
  Interventions: Dietary Supplement: VSL#3
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: VSL#3 — Dietary Supplement
  Arms: Probiotic VSL#3
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study investigates the efficacy of probiotic VSL#3 as an add on standard care on the activity of the disease in patients with Juvenile Idiopathic Arthritis.

DETAILED DESCRIPTION:
Juvenile Idiopathic Arthritis (JIA) is the most frequent rheumatic disorder in children. Numerous studies suggest that alteration of the intestinal barrier may induce abnormal immune responses implicated in development or persistence of arthritis. This paves the way to new therapeutic options aiming to reestablish intestinal homeostasis to treat arthritis or to prevent disease flares. This study investigates the efficacy of probiotic VSL#3 as an add on standard care on the activity of the disease in patients with Juvenile Idiopathic Arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥1year and <7years
* Patients with oligoarthritis and polyarthritis with rheumafactor negative and antinuclear antibodies (ANA) positive JIA with onset before the age of 6 years

Exclusion Criteria:

* Change of JIA forme

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2022-09-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of a regular intake of probiotic VSL#3 in addition to standard treatment in patients with JIA on the clinical activity | 3 months
  American College of Rheumatology Pédiatrique score (ACR Pedi )

SECONDARY OUTCOMES:
To evaluate the impact of a regular intake of probiotic VSL#3 in addition to standard treatment in patients with JIA on the intestinal microbiota. | 3 months
  Stool samples for intestinal microbiota analyses

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Meinzer, MD/PhD, Principal Investigator — APHP
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No